CLINICAL TRIAL: NCT07082361
Title: The Use of Diaphragmatic Ultrasonography: Does It Change Mechanical Ventilation Weaning Decision and Predict Outcome in COPD Patient?
Brief Title: The Use of Diaphragmatic Ultrasonography in Mechanical Ventilation Weaning Decision in COPD Patient
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shimaa Adel Mohamed Helmy Badr, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 36264MS719/10/24
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-10

CONDITIONS: Ultrasonography; Mechanical Ventilation Weaning; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Ultrasonography; Diaphragmatic; Mechanical Ventilation; Weaning
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional clinical criteria of weaning from mechanical ventilation by using spontaneous breathing (Experimental): Patients will be weaned after fulfilling the conventional clinical criteria of weaning from mechanical ventilation by using spontaneous breathing trials
  Interventions: Diagnostic Test: conventional clinical criteria and ultrasonic criteria for weaning
- conventional clinical criteria and ultrasonic criteria for weaning (Experimental): Patients will be weaned using the conventional clinical criteria and ultrasonic criteria for weaning.
  Interventions: Diagnostic Test: conventional clinical criteria of weaning from mechanical ventilation

INTERVENTIONS:
Diagnostic Test: conventional clinical criteria of weaning from mechanical ventilation — Patients will be weaned after fulfilling the conventional clinical criteria of weaning from mechanical ventilation by using spontaneous breathing trials
  Arms: conventional clinical criteria and ultrasonic criteria for weaning
Diagnostic Test: conventional clinical criteria and ultrasonic criteria for weaning — Patients will be weaned using the conventional clinical criteria and ultrasonic criteria for weaning.
  Arms: conventional clinical criteria of weaning from mechanical ventilation by using spontaneous breathing

SUMMARY:
The aim of this study is to evaluate the use of diaphragmatic ultrasonography in taking mechanical ventilation weaning decision and predicting outcome in Chronic obstructive pulmonary disease patient.

Primary outcome:

• Number of patients with failed weaning trial and need reintubation.

Secondary outcomes:

* Time till extubation trial.
* Ventilation free days after extubation less or more than 48h .
* Number of Intensive care unit discharges.
* Sensitivity and specificity of diaphragmatic assessment as a predictor of weaning.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is the fourth killer among all diseases worldwide. It can be prevented and treated, so it is an important public health challenge. Inspiratory muscle weakness has a great clinical association with Chronic obstructive pulmonary disease patients. The prolonged mechanical ventilation and weaning failure may be related to diaphragmatic muscle dysfunction. The traditional weaning parameters (e.g., spontaneous tidal volume ), Maximum inspiratory pressure , and rapid shallow breathing index are considered useful parameters for weaning. Although, they have unsatisfactory prediction rates.

Exacerbation of Chronic obstructive pulmonary disease is an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough and/or sputum beyond day-to-day variability sufficient to warrant a change in management .

In most patients, mechanical ventilation can be discontinued as soon as the underlying reason for acute respiratory failure has been resolved. However, Patients spend receiving mechanical ventilation is devoted to weaning and increase up to, 59% in Chronic obstructive pulmonary disease patients .

There are innumerable factors responsible for the failure of weaning from mechanical ventilation. Factors that should be considered in all patients include misadjusted ventilator settings, infections, airway patency and respiratory muscle performance. Malnutrition, which is common in ventilator dependent patients, has detrimental effects on the respiratory system. Heart failure or coronary ischemia can be induced by the reduction of ventilatory support which causes weaning failure. A number of electrolyte imbalances and psychological problems can be an impediment to successful weaning.

Diaphragmatic ultrasound is non-invasive, radiation-free, widely available, provides immediate and accurate results, and can be repeated at the bedside . Diaphragm sonography values provide useful information for assessing and monitoring mechanically ventilated patients .

The aim of this study is to evaluate the use of diaphragmatic ultrasonography in taking mechanical ventilation weaning decision and predicting outcome in Chronic obstructive pulmonary disease patient.

A randomized controlled study will be carried out on patients admitted to Anesthesia & Surgical intensive care unit Department in Tanta University Hospitals over a period of 1 year

ELIGIBILITY:
Inclusion Criteria:

* Adult patient more than 21 years old of both sexes, coming to our intensive care unit with acute exacerbation of Chronic obstructive pulmonary disease & need mechanical ventilation at least 48 hr.

Exclusion Criteria:

* Patient refusal.

  * Morbid obesity with body mass index > 35 kg/m2.
  * Patients with a history of recent thoracic surgery.
  * Neuromuscular disorders affecting the diaphragm e.g.(myopathy).
  * Congenital diaphragmatic disorders (Hiatal hernia).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with failed weaning trial | 28 day

SECONDARY OUTCOMES:
Time till extubation trial. | 28 days
Number of Intensive care unit discharges | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol